CLINICAL TRIAL: NCT06589570
Title: Intelligibility and Acoustic Speech Performance of CAD/CAM Milled Titanium Partial Dentures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Shady El Naggar, Principal Investigator, Badr University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-3
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Speech; Denture, Partial, Removable; CAD-CAM
MeSH Terms: conditions — Speech | interventions — Denture, Partial, Removable

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional impression-based fabrication of cobalt-chromium framework (Active Comparator): The conventional impression-based fabrication of a cobalt-chromium framework for partial dentures follows a well-established process that involves multiple steps to ensure an accurate and functional prosthesis. This method, which has been widely used for decades, relies on manual techniques and skilled craftsmanship to create the metal framework that supports the artificial teeth and secures the denture in place.
  Interventions: Device: Removable Partial Denture
- CAD design, and CAM milling of titanium framework (Experimental): The CAD (Computer-Aided Design) and CAM (Computer-Aided Manufacturing) process for creating a titanium framework for partial dentures represents a modern, highly precise approach to dental prosthesis fabrication. This digital process offers several advantages over traditional methods, such as improved accuracy, a more comfortable fit, and a reduction in the number of manual steps involved.
  Interventions: Device: Removable Partial Denture

INTERVENTIONS:
Device: Removable Partial Denture — A removable partial denture (RPD) is a dental prosthesis designed to replace one or more missing teeth in the mouth. Unlike full dentures, which are used when all teeth are missing, an RPD is specifically made for patients who still have some of their natural teeth remaining. It restores both function and aesthetics, allowing patients to chew, speak, and smile with greater confidence.

SUMMARY:
Partial dentures play a crucial role in restoring oral function and aesthetics for patients with missing teeth. Traditionally, these prostheses have been fabricated using materials such as acrylic resin or cobalt-chromium alloys. However, advancements in digital dentistry have introduced new materials and manufacturing techniques, including computer-aided design and computer-aided manufacturing (CAD/CAM) milled titanium. While titanium offers advantages such as biocompatibility, lightweight properties, and corrosion resistance, its impact on speech performance remains understudied.

DETAILED DESCRIPTION:
While the benefits of titanium in terms of durability, comfort, and biocompatibility are well-established, its impact on speech performance remains a relatively understudied aspect of its use in partial dentures. Speech is a complex function that involves the coordination of the teeth, tongue, lips, and other oral structures. The introduction of any foreign object, such as a denture, into the mouth has the potential to affect the way sounds are produced and articulated, which is why the impact of denture materials on speech must be carefully considered.

Traditional denture materials, such as acrylic resin and cobalt-chromium alloys, have been extensively studied in terms of their effects on speech performance. Research has shown that the thickness, weight, and positioning of dentures can influence how well patients are able to articulate certain sounds, particularly sibilants (such as "s" and "z" sounds) and fricatives (such as "f" and "v" sounds). Thicker or poorly fitted dentures can interfere with the movement of the tongue and lips, leading to speech distortions or difficulties in pronunciation.

Given that titanium is lighter and thinner than many traditional materials, it is reasonable to hypothesize that it could offer advantages in terms of speech performance. The reduced weight of titanium partial dentures may allow for more natural tongue and lip movements, potentially resulting in clearer and more accurate speech. Additionally, the precision of CAD/CAM technology allows for the creation of dentures that fit more snugly and comfortably in the mouth, further reducing the likelihood of speech impediments.

However, despite these potential benefits, there is currently limited research specifically focused on the impact of titanium partial dentures on speech performance. Most studies on the material have concentrated on its mechanical properties, such as strength, durability, and biocompatibility, while its effects on speech have received less attention. As speech is a vital function for communication and quality of life, further research is needed to determine whether titanium dentures offer significant improvements over traditional materials in this regard.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Class IV Kennedy Classification partial edentulism.
* Sufficient occluso-gingival height of its clinical crown
* Full opposing arch or restored with acceptable restoration
* Edentulous ridge covered by healthy firm muco-periosteum
* The abutment teeth had apparently good periodontal condition
* Adequate inter-arch space
* All patients were apparently in good general health
* Only patients who can be easily motivated to achieve and maintain good oral hygiene were selected

Exclusion Criteria:

* without abnormal bony irregularity or sever lingual undercut
* with no signs of mobility or inflammation with no tissue undercut
* Patients with shallow floor of the mouth, prominent lingual tori, bony undercuts and lingual inclined teeth were all excluded
* no tempro-mandibular joint disorders
* free from systemic diseases as diabetes mellitus

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Speech analysis | after 1 and 3 months
  Speech analysis refers to the systematic study and evaluation of human speech to understand various characteristics and functions related to sound production, articulation, and language. It is used in a wide range of fields, from linguistics and phonetics to medical and technological applications, such as diagnosing speech disorders and developing voice recognition systems.

SECONDARY OUTCOMES:
Intelligibility test | after 1 and 3 months
  An intelligibility test of speech is a method used to assess how well a person's speech is understood by others. It measures the clarity, precision, and comprehensibility of spoken words, focusing on how accurately listeners can interpret the speech without needing context or prior knowledge of the speaker's intent. Intelligibility tests are particularly important in diagnosing and evaluating speech disorders, assessing the effectiveness of speech treatments, and analyzing the impact of devices like dentures or hearing aids on communication.

CONTACTS AND LOCATIONS:
Locations (1):
- NRC, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No